CLINICAL TRIAL: NCT01454388
Title: A Randomized Controlled Trial Comparing Breakfast Versus no Breakfast
Brief Title: A Trial Comparing Breakfast Versus no Breakfast Prior to Colonoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: Hotel Dieu Hospital (Other)
Responsible Party: Principal Investigator, Dr. Lawrence Hookey, Principal Investigator, Queen's University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: breakfast colonoscopy study
Record Dates: First submitted 2011-10-12; First posted 2011-10-19 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Clinically Indicated Colonoscopy
MeSH Terms: interventions — Breakfast

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- PEG plus breakfast (Active Comparator): patients are allowed to have a low residue breakfast the day prior to colonoscopy
  Interventions: Other: breakfast
- PEG without breakfast (No Intervention)
- picosalax plus breakfast (Active Comparator): patients are allowed to have a low residue breakfast the day prior to colonoscopy
  Interventions: Other: breakfast
- picosalax without breakfast (No Intervention)

INTERVENTIONS:
Other: breakfast
  Arms: PEG plus breakfast; picosalax plus breakfast

SUMMARY:
In addition to bowel cleansing agents, the current practice of bowel preparation for colonoscopy involves a low residue diet 48 hours prior to and a clear fluid diet the day before the procedure. This study aims to test whether patients who consume a low residue breakfast the day prior to colonoscopy have a difference in the quality of their bowel preparation. Patients requiring outpatient colonoscopies will be asked to participate. They will be randomized to either breakfast or no breakfast the day before the procedure. Colon cleanliness, patient hunger, and tolerance will be assessed.

The investigators hypothesize that there will be no difference in bowel preparation scores and will be better tolerated

DETAILED DESCRIPTION:
Colon cleansing prior to colonoscopy is essential for an adequate examination. Research has shown that preparation prior to colonoscopy remains one of the biggest deterrents for patients considering colon screening (1).

In addition to the bowel cleansing agents another important aspect of the preparation is the diet consumed prior to the procedure. Currently 48 hours prior to colonoscopy patients are asked to consume a low residue diet. The day before the procedure they are switched to a clear fluid only diet which many patients find difficult to follow due to hunger and can lead to non-compliance with the preparation.

There have been no trials to date which have answered the question whether the consumption of breakfast alters colon cleansing with the cleansing agents currently used in Canada. Investigators found that in patients receiving sodium phosphate preparations, a full breakfast or low residue lunch had no effect on colon cleansing scores and improved hunger and energy levels (2). Several studies have looked at the result of low residue diet kits taken the day prior to the procedure and showed no difference in colon cleansing or tolerability compared to the traditional clear fluid regime (3,4).

This study aims to test whether patients who consume a low residue breakfast the day prior to colonoscopy have a difference in the quality of their colon cleansing or tolerability of the preparation compared to those who consume a clear fluid diet. The investigators hypothesize that there will be no difference in bowel preparation scores and will be better tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Patients for whom a GI physician has ordered a colonoscopy will be approached for inclusion in the trial

Exclusion Criteria:

* ileus or bowel obstruction -significant constipation (<3 spontaneous bowel movements/day)- previous colorectal surgery
* ascites
* active inflammatory bowel disease
* pregnancy
* recent (<6 months) myocardial infarction or unstable angina

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 496 (Actual)
Dates: Start 2010-01; Primary Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
bowel cleansing efficacy | 2 days
  Quality of bowel cleansing as measured by Ottawa Bowel Scale

SECONDARY OUTCOMES:
Hunger | day of colonoscopy (day 1)
  Using a tolerance scale and VAS hunger will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Hookey, MD, Principal Investigator — Queen's University
Locations (1):
- Hotel Dieu Hospital, Kingston, Ontario, Canada

REFERENCES:
- [Derived] Flemming JA, Green J, Melicharkova A, Vanner S, Hookey L. Low-residue breakfast during the preparation for colonoscopy using a polyethylene glycol electrolyte solution: a randomised non-inferiority trial. BMJ Open Gastroenterol. 2015 May 28;2(1):e000029. doi: 10.1136/bmjgast-2015-000029. eCollection 2015. PMID 26462280